CLINICAL TRIAL: NCT03420872
Title: Prenatal and Childhood Nutrient Mixtures Predict Neurodevelopmental Outcomes Among Children in Mexico City
Brief Title: Nutrient Mixtures and Neurodevelopment
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 12-1417
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Neurodevelopment
Keywords: Nutrition; Nutrients; Mixtures; Neurodevelopment; Prenatal; Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subset from PROGRESS cohort: Participants included children 4-6 years of age from mother-child pairs in the Programming Research in Obesity, Growth Environment and Social Stress (PROGRESS) prospective birth cohort in Mexico City
  Interventions: Other: Nutrient mixtures

INTERVENTIONS:
Other: Nutrient mixtures — consumption of a mixture of beneficial nutrients

SUMMARY:
Background: Adequate levels of beneficial nutrients are important for neurodevelopment. Although, nutrients are ingested in combination, considering nutrients as a mixture has not been studied with respect to health, such as neurodevelopment.

Objective: To examine the impact of prenatal and childhood nutrition mixtures on neurodevelopment.

Design: Participants included mother-child pairs in the Programming Research in Obesity, Growth Environment and Social Stress (PROGRESS) prospective birth cohort in Mexico City. Prenatal and child nutrition profiles were assessed among 65 and 329 children respectively by analyzing components of a food frequency questionnaire. Child neurodevelopmental outcomes at 4-6 years of age were measured using the McCarthy Scales of Children's Abilities (MSCA).

ELIGIBILITY:
Inclusion Criteria:

Women of children:

* less than 20 weeks gestation at the start of the study
* at least 18 years of age
* and planned to reside in Mexico City for the next three years.

Exclusion Criteria:

Women of children:

* free of heart or kidney disease
* not use steroids or anti-epilepsy drugs
* not consume alcohol.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy pregnant women living in Mexico city from 2006-2009 seeking health care in clinics (Parent-child pairs) and their children at 4 - 6 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2006-09-15 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
McCarthy Scales of Children's Abilities (MSCA) | at age 4
  The MSCA consists of 18 short sub-tests that are weighted and combined to yield five scale scores or indexes - verbal, perceptual performance, quantitative, memory and motor - as well as an overall general cognitive index based on the first three scaled indexes. The McCarthy Scale index scores can range from 22 - 78 with higher index scores indicating better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wright, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai; Mara Tellez-Rojo, PhD, Principal Investigator — National Institute of Public Health, Mexico
Locations (1):
- National Institute of Public Health, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Munoz-Rocha TV, Tamayo Y Ortiz M, Romero M, Pantic I, Schnaas L, Bellinger D, Claus-Henn B, Wright R, Wright RO, Tellez-Rojo MM. Prenatal co-exposure to manganese and depression and 24-months neurodevelopment. Neurotoxicology. 2018 Jan;64:134-141. doi: 10.1016/j.neuro.2017.07.007. Epub 2017 Jul 17. PMID 28728787
- [Background] Rodosthenous RS, Burris HH, Svensson K, Amarasiriwardena CJ, Cantoral A, Schnaas L, Mercado-Garcia A, Coull BA, Wright RO, Tellez-Rojo MM, Baccarelli AA. Prenatal lead exposure and fetal growth: Smaller infants have heightened susceptibility. Environ Int. 2017 Feb;99:228-233. doi: 10.1016/j.envint.2016.11.023. Epub 2016 Dec 5. PMID 27923585
- [Background] Rosa MJ, Just AC, Guerra MS, Kloog I, Hsu HL, Brennan KJ, Garcia AM, Coull B, Wright RJ, Tellez Rojo MM, Baccarelli AA, Wright RO. Identifying sensitive windows for prenatal particulate air pollution exposure and mitochondrial DNA content in cord blood. Environ Int. 2017 Jan;98:198-203. doi: 10.1016/j.envint.2016.11.007. Epub 2016 Nov 11. PMID 27843010
- [Background] Renzetti S, Just AC, Burris HH, Oken E, Amarasiriwardena C, Svensson K, Mercado-Garcia A, Cantoral A, Schnaas L, Baccarelli AA, Wright RO, Tellez-Rojo MM. The association of lead exposure during pregnancy and childhood anthropometry in the Mexican PROGRESS cohort. Environ Res. 2017 Jan;152:226-232. doi: 10.1016/j.envres.2016.10.014. Epub 2016 Oct 28. PMID 27810680
- [Background] Burris HH, Baccarelli AA, Byun HM, Cantoral A, Just AC, Pantic I, Solano-Gonzalez M, Svensson K, Tamayo y Ortiz M, Zhao Y, Wright RO, Tellez-Rojo MM. Offspring DNA methylation of the aryl-hydrocarbon receptor repressor gene is associated with maternal BMI, gestational age, and birth weight. Epigenetics. 2015;10(10):913-21. doi: 10.1080/15592294.2015.1078963. Epub 2015 Aug 7. PMID 26252179
- [Background] Sanders AP, Burris HH, Just AC, Motta V, Svensson K, Mercado-Garcia A, Pantic I, Schwartz J, Tellez-Rojo MM, Wright RO, Baccarelli AA. microRNA expression in the cervix during pregnancy is associated with length of gestation. Epigenetics. 2015;10(3):221-8. doi: 10.1080/15592294.2015.1006498. PMID 25611922